CLINICAL TRIAL: NCT02007265
Title: Post-stroke Triage "DOC": Simple Screening for Depression, Obstructive Sleep Apnea and Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Dr. Richard H. Swartz, Dr. Richard Swartz, Sunnybrook Health Sciences Centre
Other Study IDs: 306-2011; No. 000392 (Other Grant/Funding Number: Heart and Stroke Foundation of Ontario Grant)
Record Dates: First submitted 2013-11-13; First posted 2013-12-10 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Transient Ischemic Attack; Stroke; Depression; Obstructive Sleep Apnea; Cognitive Impairment
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke; Depression; Sleep Apnea, Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TIA and SPC outpatients: All consecutive patients attending outpatient TIA and Stroke Prevention Clinics at three regional stroke centres will be eligible to be screened.

SUMMARY:
The purpose of this study is to determine whether simple, evidence-based clinical screening be quickly and feasibly implemented (>85% of patients in an average of <6 minutes) in large-volume urgent transient ischemic attack (TIA)/stroke clinics to identify individuals at high risk for the three most common and devastating post-stroke co-morbidities (depression, obstructive sleep apnea and cognitive disorders).

DETAILED DESCRIPTION:
We have created a simple screening tool (the "DOC" Screen) that will be routinely applied to all patients at a high-volume Regional Stroke Prevention Clinic. Consenting patients will also undergo "gold standard" research assessments in order to determine the diagnostic characteristics of the screen compared to gold standard research assessments.The proportion of eligible patients who complete DOC screening and the time for completion (mean, range, standard deviations) will be calculated from aggregated data for all new consults in the stroke prevention clinic. For patients who consented to undergo gold standard testing, sensitivity, specificity, positive predictive value, negative predictive value and likelihood ratios of the DOC screen will be calculated. Screening cut-points will be optimized using Receiver Operating Characteristic (ROC) and area under the curve analysis, and logistic regression will be applied to this ROC Curve analysis to control for variables such as age, sex, BMI and education. We hope to develop a pragmatic approach to screening the large, high-risk stroke prevention clinic population, allowing broad screening for these important health conditions. This could change routine standard of care across stroke prevention clinics and facilitate early identification and appropriate assessment of patients.

ELIGIBILITY:
Inclusion Criteria:

* Attending outpatient TIA and Stroke Prevention Clinics at any of the three regional stroke centres.

Exclusion Criteria:

* Those who are unable to complete the screen complete the screen due to severe aphasia, severe motor dysfunction and those who are not fluent in English without translation available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients attending outpatient TIA and Stroke Prevention Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1504 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with who completed the DOC Screen in 5 minutes or less | Day 1
  This outcome is defined as the number of DOC patients that took 5 minutes or less to complete the DOC Screening Form

SECONDARY OUTCOMES:
DOC Screen Diagnostic Characteristics compared to Gold Standard Research Assessments | Average 7 weeks
  To determine the diagnostic characteristics of the mini-screens compared to gold standard research assessments and to determine whether when applied as one integrated test in a stroke clinic population they perform comparably to previously published studies.

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Swartz, MD, PhD,, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada